CLINICAL TRIAL: NCT01411150
Title: Premanifest Huntington's Disease: Creatine Safety & Tolerability Extension Study
Acronym: Pre-CREST-X
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Steven M. Hersch, Professor of Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000642
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Huntington's Disease
Keywords: Premanifest; At-Risk; Huntington's Disease; HD
MeSH Terms: conditions — Huntington Disease | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Creatine (Experimental)
  Interventions: Drug: Creatine Monohydrate

INTERVENTIONS:
Drug: Creatine Monohydrate — Up to 30 grams daily creatine monohydrate

SUMMARY:
The purpose of this clinical trial is to extend the Pre-Crest study (Protocol # (NCT00592995) to further assess the long-term safety and tolerability of up to 30 grams daily creatine in individuals at-risk for Huntington's Disease (HD) and to assess whether biomarkers responsive to creatine in symptomatic individuals are informative in premanifest individuals over a longer duration.

DETAILED DESCRIPTION:
Extensive evidence exists that neurodegeneration begins many years before HD can be diagnosed clinically. Therefore, it is most desirable to begin a neuroprotective therapy before or during this premanifest period with the aim of delaying onset, as well as slowing functional decline. Cellular energy depletion is present early in HD and can be ameliorated by creatine, which helps regenerate cellular ATP. Preclinical evidence for creatine's potential neuroprotective effects in animal models of HD has been well-documented. Before the clinical efficacy of creatine can be tested in premanifest HD, its long-term safety and tolerability must be assessed in these individuals and its ability to favorably modify biomarkers of HD should also be confirmed. This extension trial will continue to follow eligible individuals who completed the PreCREST study on open-label creatine (up to 30 grams daily) for long term safety and tolerability. Additional biological and imaging biomarkers of disease progression and potential response to treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have completed the Pre-CREST Study.
* Individuals capable of providing independent informed consent and complying with trial procedures.

Exclusion Criteria:

-Clinical evidence of unstable medical or psychiatric illness in the investigator's judgment.

Additional eligibility criteria apply.

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  Frequency of adverse events
Tolerability | 12 months
  Proportion of subjects completing the extension study at given dose level

SECONDARY OUTCOMES:
Clinical measures | 12 months
  Components of the UHDRS (United Huntington's Disease Rating Scale)
Biological Markers of Disease Progression | 12 Months
  Biological indicators that creatine treatment might affect the progression of HD: plasma levels of creatine, serum levels of 8OH2'dG and 8OHG, magnetic resonance imaging (MRI), morphometric neuroimaging (biomarker of neurodegeneration), metabolomic profiling, and gene expression analysis to assess transcriptional effects of HD and creatine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Rosas, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Background] Rosas HD, Reuter M, Doros G, Lee SY, Triggs T, Malarick K, Fischl B, Salat DH, Hersch SM. A tale of two factors: what determines the rate of progression in Huntington's disease? A longitudinal MRI study. Mov Disord. 2011 Aug 1;26(9):1691-7. doi: 10.1002/mds.23762. Epub 2011 May 24. PMID 21611979
- [Background] Kim J, Amante DJ, Moody JP, Edgerly CK, Bordiuk OL, Smith K, Matson SA, Matson WR, Scherzer CR, Rosas HD, Hersch SM, Ferrante RJ. Reduced creatine kinase as a central and peripheral biomarker in Huntington's disease. Biochim Biophys Acta. 2010 Jul-Aug;1802(7-8):673-81. doi: 10.1016/j.bbadis.2010.05.001. Epub 2010 May 9. PMID 20460152
- [Background] Rosas HD, Lee SY, Bender AC, Zaleta AK, Vangel M, Yu P, Fischl B, Pappu V, Onorato C, Cha JH, Salat DH, Hersch SM. Altered white matter microstructure in the corpus callosum in Huntington's disease: implications for cortical "disconnection". Neuroimage. 2010 Feb 15;49(4):2995-3004. doi: 10.1016/j.neuroimage.2009.10.015. Epub 2009 Oct 19. PMID 19850138
- [Background] Rosas HD, Salat DH, Lee SY, Zaleta AK, Hevelone N, Hersch SM. Complexity and heterogeneity: what drives the ever-changing brain in Huntington's disease? Ann N Y Acad Sci. 2008 Dec;1147:196-205. doi: 10.1196/annals.1427.034. PMID 19076442
- [Background] Hersch SM, Rosas HD. Neuroprotection for Huntington's disease: ready, set, slow. Neurotherapeutics. 2008 Apr;5(2):226-36. doi: 10.1016/j.nurt.2008.01.003. PMID 18394565
- [Background] Rosas HD, Salat DH, Lee SY, Zaleta AK, Pappu V, Fischl B, Greve D, Hevelone N, Hersch SM. Cerebral cortex and the clinical expression of Huntington's disease: complexity and heterogeneity. Brain. 2008 Apr;131(Pt 4):1057-68. doi: 10.1093/brain/awn025. Epub 2008 Mar 12. PMID 18337273
- [Background] Hersch SM, Gevorkian S, Marder K, Moskowitz C, Feigin A, Cox M, Como P, Zimmerman C, Lin M, Zhang L, Ulug AM, Beal MF, Matson W, Bogdanov M, Ebbel E, Zaleta A, Kaneko Y, Jenkins B, Hevelone N, Zhang H, Yu H, Schoenfeld D, Ferrante R, Rosas HD. Creatine in Huntington disease is safe, tolerable, bioavailable in brain and reduces serum 8OH2'dG. Neurology. 2006 Jan 24;66(2):250-2. doi: 10.1212/01.wnl.0000194318.74946.b6. PMID 16434666
- [Background] Rosas HD, Tuch DS, Hevelone ND, Zaleta AK, Vangel M, Hersch SM, Salat DH. Diffusion tensor imaging in presymptomatic and early Huntington's disease: Selective white matter pathology and its relationship to clinical measures. Mov Disord. 2006 Sep;21(9):1317-25. doi: 10.1002/mds.20979. PMID 16755582
- [Background] Ryu H, Rosas HD, Hersch SM, Ferrante RJ. The therapeutic role of creatine in Huntington's disease. Pharmacol Ther. 2005 Nov;108(2):193-207. doi: 10.1016/j.pharmthera.2005.04.008. Epub 2005 Aug 1. PMID 16055197
- [Background] Borovecki F, Lovrecic L, Zhou J, Jeong H, Then F, Rosas HD, Hersch SM, Hogarth P, Bouzou B, Jensen RV, Krainc D. Genome-wide expression profiling of human blood reveals biomarkers for Huntington's disease. Proc Natl Acad Sci U S A. 2005 Aug 2;102(31):11023-8. doi: 10.1073/pnas.0504921102. Epub 2005 Jul 25. PMID 16043692
- [Background] Rosas HD, Liu AK, Hersch S, Glessner M, Ferrante RJ, Salat DH, van der Kouwe A, Jenkins BG, Dale AM, Fischl B. Regional and progressive thinning of the cortical ribbon in Huntington's disease. Neurology. 2002 Mar 12;58(5):695-701. doi: 10.1212/wnl.58.5.695. PMID 11889230
- [Background] Hersch SM, Rosas HD. Neuroprotective therapy for Huntington's disease: new prospects and challenges. Expert Rev Neurother. 2001 Sep;1(1):111-8. doi: 10.1586/14737175.1.1.111. PMID 19811052
- [Background] Stack EC, Dedeoglu A, Smith KM, Cormier K, Kubilus JK, Bogdanov M, Matson WR, Yang L, Jenkins BG, Luthi-Carter R, Kowall NW, Hersch SM, Beal MF, Ferrante RJ. Neuroprotective effects of synaptic modulation in Huntington's disease R6/2 mice. J Neurosci. 2007 Nov 21;27(47):12908-15. doi: 10.1523/JNEUROSCI.4318-07.2007. PMID 18032664
- [Background] Dedeoglu A, Kubilus JK, Yang L, Ferrante KL, Hersch SM, Beal MF, Ferrante RJ. Creatine therapy provides neuroprotection after onset of clinical symptoms in Huntington's disease transgenic mice. J Neurochem. 2003 Jun;85(6):1359-67. doi: 10.1046/j.1471-4159.2003.01706.x. PMID 12787055